CLINICAL TRIAL: NCT03237507
Title: Prospective and Non-interventional Study on Peritoneal Metastasis of Stage IV Gastric Cancer
Brief Title: Nonintervention Study on Peritoneal Metastasis of Stage IV Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Wang Kuan, M.D.Prof, Professor, Harbin Medical University
Other Study IDs: TOTPMSG1602
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Stage IV Gastric Cancer With Metastasis
MeSH Terms: interventions — S 1 (combination); Oxaliplatin; Hyperthermic Intraperitoneal Chemotherapy; Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy Group: chemotherapy treatment（S-1 and Oxaliplatin） for patients until disease progress
  Interventions: Drug: S-1; Drug: oxaliplatin
- Chemotherapy plus HIPEC Group: Hyperthermic Intraperitoneal chemoperfusion（HIPEC）with Paclitaxel more than 2 cycles and plus chemotherapy
  Interventions: Drug: S-1; Drug: oxaliplatin; Device: Hyperthermic Intraperitoneal; Drug: Paclitaxel

INTERVENTIONS:
Drug: S-1 — 40-60mg/m^2 bid, days 1-14, oral，every 3 weeks.
Drug: oxaliplatin — 100mg/m^2 days 1，intravenous infusion, every 3 weeks.
Device: Hyperthermic Intraperitoneal — hyperthermic intraperitoneal chemoperfusion
  Groups: Chemotherapy plus HIPEC Group
Drug: Paclitaxel — intraperitoneal perfusion
  Groups: Chemotherapy plus HIPEC Group

SUMMARY:
This is a non-interventional study，aim to observe the safety and efficiency of different treatment regimen for peritoneal metastasis of Stage IV gastric cancer in the real world

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age
* Patients with histologically confirmed gastric cancer or gastroesophageal junction adenocarcinoma, stage IV with peritoneal metastasis
* Didn't received any prior systemic chemotherapy
* Signed informed consent

Exclusion Criteria:

* History of hypersensitivity to fluoropyrimidines, Tegafur，Gimeracil and Oteracil Potassium Capsules , capecitabine, oxaliplatin or the ingredients of this product
* Pregnancy or lactation women,
* Inadequate hematopoietic function： WBC≦3,500/mm3; ANC≦1,500/mm3; Platelet≦80,000/mm3
* Inadequate organ function which is defined as below:

Total bilirubin >2 pper limit of normal range (ULN); ALT / AST > 2.5 upper limit of normal range (ULN); serum creatinine > 1.5 mg/dL, and Ccr > 60 ml/min (estimated by Cockcroft-Gault formulation);

* Symptomatic peripheral neuropathy
* Receiving a concomitant treatment with other fluoropyrimidines
* Fluoropyrimidines (DPD) congenital absence
* Other Situations which physicians suggesting are inadaptable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed gastric cancer or gastroesophageal junction adenocarcinoma, stage IV with peritoneal metastasis
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS: Progression Free Survival | through study completion, an average of 1 year
  time from enrollment to disease progression or death

SECONDARY OUTCOMES:
OS:overall survival | 3 years
  time from enrollment to death
Safety | 3 years
  measured by recording the subjects' Adverse Events according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Kuan Wang, Principal Investigator — Harbin Medical University Cancer Hospital,Gastrointestinal Surgical department
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China